CLINICAL TRIAL: NCT06398379
Title: Virus as Treatment of C. Difficile Infection (VISION)
Acronym: VISION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Frederik Cold, MD, PhD, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-22069168
Record Dates: First submitted 2024-03-21; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Clostridium Difficile Infections
Keywords: Fecal Virome Transplantation; Fecal Microbiota Transplantation
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial comparing study treatment (Fecal Virome Transplantation) to standard treatment (Fecal Microbiota Transplantation)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Fecal Virome Transplantation and Fecal Microbiota Transplantation capsules will look exactly the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Virome Transplantation (Experimental): Treatment with Fecal Virome Transplantation capsules (one treatment) following standard treatment of antiobiotics (Vancomycin)
  Interventions: Other: Fecal Virome Transplantation
- Fecal Microbiota Transplantation (Active Comparator): Treatment with Fecal Microbiota Transplantation capsules (one treatment) following standard treatment of antiobiotics (Vancomycin)
  Interventions: Other: Fecal microbiota Transplantation

INTERVENTIONS:
Other: Fecal Virome Transplantation — The primary steps of the production of fecal virome transplantation capsules is the same as when producing fecal microbiota transplantation capsules. Through an subsequent proces of filtering bacterial parts of the material are removed. The material, now called fecal virome transplanation material, has then been moved to capsules and stored in -80c untill use.
  Other Names: Sterile fecal filtrate
  Arms: Fecal Virome Transplantation
Other: Fecal microbiota Transplantation — Donor fecal material is mixed with cryoprotectant and NaCl. Following processing the material transfered to capsules and is stored at -80c prior to use.
  Other Names: FMT
  Arms: Fecal Microbiota Transplantation

SUMMARY:
Fecal Virome Transplantation (FVT) has in small studies shown benefit in the treatment of recurrent C. difficile infection.

In the VISION study we will treat patients with recurrent C. difficile infection with FVT capsules and compare the treatment with Fecal Microbiota Transplantation (FMT) capsules. Both will be following af standard treatment of antibiotics (Vancomycin)

DETAILED DESCRIPTION:
In the VISION study we will treat patients with recurrent C. difficile infection (CDI) with FVT capsules and compare the treatment with Fecal Microbiota Transplantation (FMT) capsules. Patients will be randomised to receive either FMT or FTV capsules.

Patients will be followed for one year to investigate the risk of a new recurrence of CDI.

Patients and researchers involved in the treatment of the patients will be blinded to the treatment

ELIGIBILITY:
Inclusion Criteria:

* Recurrent C. difficile infection (first or second recurrence)
* Understand danish

Exclusion Criteria:

* Serious food allergy (anaphylaxis)
* Other pathogenic bacteria/virus in stool sample prior to inclusion
* Inability to ingest capsules
* Gastrointestinal perforation in the 180 days prior to inclusion
* Previous treatment with FMT og rectal bacteriotherapy in the 180 days prior to inclusion
* Short bowel syndrome
* Pregnancy or planning of pregnancy
* Participation in other clinical trial in the 30 days prior to inclusion
* Stoma
* Other condition where FMT is considered contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical resolution (≤ 3 bowel movements) or diarrhoea with a negative stool sample for C. diffiicile) | 8 weeks following treatment
  Number of patients in each group (FMT and FVT) with clinical resolution
Participation | 1 week after given information about the study
  Among patients eligible for treatment how many are interesting in participating in study and potentially receiving new virome treatment

SECONDARY OUTCOMES:
Need for rescue Fecal Microbiota Transplantation (FMT) | Up til eight weeks following treatment
  Number of patients with diarrhoea and stool sample positive for C. diffiicile needing rescue-FMT
Long term recurrence of C. difficile infection | Up to one year following treatment
  Number of patients registered with recurrence of C. difficile infection (through a positive stool sample) in the first year following treatment
Side effects | Up to eight weeks following treatment
  Registered side effects in the first 8 weeks following treatment

OTHER OUTCOMES:
Microbiome changes | Through samples prior to treatment, one and eight weeks following treatment
  Microbiome changes in fecal virome and bacteriome following FMT and FVT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Cold, MD, PhD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No